CLINICAL TRIAL: NCT04867304
Title: Determinants of Depression and Its Impact on Quality of Life in Patients With Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rupjyoti Talukdar, Director, Pancreas Clinic; Head, Pancreas Research Group, Asian Institute of Gastroenterology, India
Other Study IDs: AIG-DEPCP-01
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pancreatitis; Depression; Quality of Life; Chronic Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Depression; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: Individuals without any known illnesses and normal labs./USG w/a. This group was used to compare baseline depression, magnetic resonance spectroscopy and plasma metabolites.
- Chronic pancreatitis without depression: This group contains patients with CP who does not have depression based on the Beck Depression inventory.
  Interventions: Other: Patient education about chronic pancreatitis.
- Chronic pancreatitis with depression: This group contains patients with CP who has depression based on the Beck Depression inventory.
  Interventions: Other: Patient education about chronic pancreatitis.

INTERVENTIONS:
Other: Patient education about chronic pancreatitis. — Patients in the second cohort were educated about their disease phenotype in a structured and personalised manner that included their disease course, symptoms, imaging, treatment option and possible long-term outcomes and prognosis. This was followed by answering all the queries of the patient and their caregivers.
  The patients were advised to visit the Pancreas clinic after 3-months for re-evaluation of the clinical, psychological and metabolic parameters.
  Groups: Chronic pancreatitis with depression; Chronic pancreatitis without depression

SUMMARY:
Chronic pancreatitis (CP) is associated with recurrent intractable abdominal pain, pancreatic exocrine insufficiency and endocrine dysfunction. Very few studies had evaluated the quality of life in CP, and even a fewer have assessed the mental status in these patients.

In the current study, we proposed to evaluate the the relationship between pain, quality of life and depression status in two large independent cohorts of patients with CP. We also proposed to evaluate the brain metabolites in the right and left anterior cingulate cortex, basal ganglia, hippocampus and prefrontal cortex using magnetic resonance spectroscopy. We further proposed to evaluate the pasta metabolites and look for associations with the mental state. Finally, we proposed to evaluate how CP related education of the patients could impact on their mental status and response to interventions on pain.

ELIGIBILITY:
A. Inclusion Criteria:

* Age 18-60yrs
* Both genders
* Documented CP for at least 3 years
* Capable and willing to provide informed consent

B. Exclusion Criteria:

* Acute exacerbation of pancreatitis
* Pancreatic malignancy
* On anti-depressant and antipsychotic medications
* Concomitant psychiatric illness (other than depression)
* Pancreatic malignancy
* Major co-morbidities
* Pregnancy and lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population constitutes of patients with chronic pancreatic of at least 3 years duration. They are a composite with or without depression. Rationale for taking a lag time of at least 3 years was to allow development of the complications of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement in depression scores | 3 months
  Measured by the BDI II score
Improvement in Quality of life parameters | 3 months
  Measured by the EORTC-QLQc30 + PAN28
Change in brain metabolite profiles | 3 months
  Measured by using Magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India